CLINICAL TRIAL: NCT06616038
Title: Biomarker Assessment in Heart Failure with Reduced Systolic Function (HFrEF) and Preserved Systolic Function (HFpEF)
Brief Title: Heart Failure Biomarkers
Acronym: BIOHF
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: BIOHF
Record Dates: First submitted 2024-09-18; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation (AF); Hart Failure
Keywords: Hart failure; Ejection fraction; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- heart failure patients (HFrEF and HFpEF) without atrial fibrillation: Will be enrolled 57 patients with heart failure patients (HFrEF and HFpEF) without atrial fibrillation
  Interventions: Other: Data collection
- heart failure patients (HFrEF and HFpEF) with atrial fibrillation: Will be enrolled 57 patients with heart failure patients (HFrEF and HFpEF) with atrial fibrillation
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Given the observational nature of the study, the intervention is a simple data collection

SUMMARY:
Systemic inflammation is closely associated with the development and progression of heart failure (HF). The study assessed the fibrin/albumin (FAR) ratio, a very important biomarker, as a prognostic indicator of HE. Study population is composed by patients who were addicted with heart failure diagnosed for the first time or already under treatment (NYHA class II-IV) and reduced ejection fraction (HFrEF) or preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Prospective, observational, single-center study, which involves the enrollment of patients affected by heart failure of first diagnosis or already in therapy, who will be subjected to an analysis of the Albumin/fibrinogen ratio. Subjects will not be subjected to specific visits or services for the study: clinical and anamnestic data will be collected during routine visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients with newly diagnosed or already treated heart failure (NYHA class II-IV) with HFrEF and HFpEF with and without atrial fibrillation.
* Patients who sign the consent to participate in the study

Exclusion Criteria:

* Patients with infectious/autoimmune diseases, neoplasms, liver failure, renal failure (Cl creatinine < 30 mL/L), structural cardiomyopathies and pericarditis.
* Pregnant/breastfeeding women (verified by self-declaration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be enrolled 114 patients admitted to the Hospital for heart failure of first diagnosis or already undergoing therapy. In particular, 57 patients with heart failure and 57 patients with heart failure and fibrillation will be included.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of FAR | At Hospital admission
  Evaluate FAR (=Fibrin/Albumin) in heart failure HFrEF and HFpEF with or without atrial fibrillation.

SECONDARY OUTCOMES:
FAR (=Fibrinogen/Albumin) and functional ultrasound | At Hospital admission and at hospital discharge (assessed up to 1 months)
  Correlate FAR to functional ultrasound indices of atrium and ventricle and to the presence of atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy
  - IRCCS Galeazzi-Sant'Ambrogio, Milan

IPD SHARING:
Plan to Share IPD: Undecided